CLINICAL TRIAL: NCT04547478
Title: Evaluation of Low Muscle Mass by Muscle Surface Index of First Lumbar Vertebrae Using Low Dose Computed Tomography
Brief Title: L1 M1 of LDCT for Low Muscle Mass Measurement
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-107091-E
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: low dose chest CT(LDCT) — cross sectioned muscle area of the 1st vertebrae level obtained by LDCT

SUMMARY:
The first lumbar spine muscle index (L1 MI) on computed tomography (CT) obtained by measuring muscle surface at the first lumbar vertebrae (L1) level is an indicator of total skeletal mass in specific populations. Nevertheless, the utility of L1 MI derived from low dose chest CT (LDCT) in health assessments and relevant cutoff points are unclear.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 20 years who received LDCT in routine health assessments from January to December 2017 were enrolled at a tertiary care hospital (Far Eastern Memorial Hospital, New Taipei City, Taiwan).

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects in routine health assessments
Sampling Method: Non-Probability Sample
Enrollment: 3304 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Cross sectional muscle area of the 1st vertebrae level | 52 weeks
  Cross sectional muscle area of the 1st vertebrae level by LDCT

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No